CLINICAL TRIAL: NCT04015180
Title: An Extension Study to Evaluate the Long-term Outcomes of Subjects Who Received Treatment for Retinopathy of Prematurity in Study 20090
Brief Title: Extension Study to Evaluate the Long-term Outcomes of Subjects in Study 20090
Acronym: FIREFLEYE next
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20275; 2023-504207-89-00 (Other: CTIS (EU)); 2018-003180-54 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept arm (Experimental): No study treatment will be administered. The treatments to be evaluated in this study were administered in Study 20090.
  Interventions: Drug: Eylea (Aflibercept, BAY86-5321)
- Laser photocoagulation arm (Active Comparator): No study treatment will be administered. The treatments to be evaluated in this study were administered in Study 20090.
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Drug: Eylea (Aflibercept, BAY86-5321) — Treatment administered in 20090. Solution in a sterile glass vial, Dose A, IVT injection.
  Arms: Aflibercept arm
Procedure: Laser photocoagulation — Treatment administered in 20090. Transpupillary conventional laser ablative therapy
  Arms: Laser photocoagulation arm

SUMMARY:
This is a follow-up study to evaluate the long term outcome of babies treated in the FIREFLEYE study.

ELIGIBILITY:
Inclusion Criteria:

* Subject was treated in Study 20090
* Age less than 13 months of chronological age
* Signed informed consent from parent(s)/legally authorized representative(s), which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

- Subject has a condition preventing participation in the study, or performance of study procedures.

Max Age: 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Binocular best-corrected visual acuity in Snellen equivalent | At 5 years of age.
Proportion of subjects with ocular AEs and SAEs | Up to 5 years of age.
  AE: adverse event SAE: serious adverse event
Proportion of subjects with systemic AEs and SAEs | Up to 5 years of age.

SECONDARY OUTCOMES:
Proportion of subjects developing unfavorable ocular structural outcome | At 1,3 and 5 years of age.
  Unfavorable ocular structural outcome include:
  retinal detachment, macular dragging, macular fold, retrolental opacity
Proportion of subjects with absence of active ROP and unfavorable structural outcomes | At 1 year of age.
Best-corrected visual acuity in each eye | At 3 and 5 years of age.
Refractive spherical equivalent in each eye | At 3 and 5 years of age
Neurodevelopmental outcomes using BSID-III | At 2 years of age
  BSID-III: The Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) is a standard series of tests that will assess the development of children in 3 areas: cognition, language, and motor skills. It is recommended to be assessed at screening, 1 year and 2 years of age. The assessment at 2 years of age is mandatory.
Neurodevelopmental outcomes using WPPSI-IV | At 5 years of age
  WPPSI-IV: The Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition is designed to assess development of older children and is recommended to be performed at 3, 4 and 5 years of age. The assessment at 5 years of age is mandatory. In cases where the WPSSI-IV cannot be used, the Differential Ability Scales II (DAS-II) may be used as an alternative.
Neurodevelopmental outcomes using VABS-II | At 2 and 5 years of age
  VABS-II: Vineland Adaptive Behavior Scales, Second Edition Expanded Interview will be included, which includes 4 areas: Communication, Daily Living skills, Socialization and Motor Skills. It is recommended to be assessed at 2, 3, 4 and 5 years of age. The assessments at 2 years and 5 years of age are mandatory.
Proportion of subjects with recurrence of ROP | At 3 and 5 years of age.
Proportion of subjects requiring treatment for ROP | Up to 5 years of age.
Proportion of subjects requiring ophthalmological treatment | Up to 5 years of age.

CONTACTS AND LOCATIONS:
Locations (55):
- Hospital Público Descentralizado "Dr. Guillermo Rawson", San Juan, Argentina
- AZ Sint Jan Brugge - Ophthalmology, Bruges, Belgium
- Brazil (2):
  - Hospital das Clínicas de Botucatu - UNESP Botucatu, Botucatu, São Paulo
  - Unifesp/Epm, São Paulo
- Bulgaria (4):
  - UMHAT Sveti Georgi, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - Spec. Hospital of Ophthalm. for Active Treatment Visus, Sofia
  - Spec. Hosp. of Ophthalm. Disease for Active Treatment Varna, Varna
- Czechia (2):
  - Fakultní nemocnice Ostrava, Ostrava
  - Všeobecná fakultní nemocnice v Praze, Prague
- Greece (3):
  - Children's Hospital of Athens P&A Kyriakou - Pediatric Nephrology Department, Athens
  - General Hospital Of Thessaloniki Papageorgiou-2nd Ophthalmology Clinic, Efkarpia
  - University General Hospital of Ioannina, Ioannina
- Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz és Szakrendelo, Budapest, Hungary
- Kaplan Medical Center, Rehovot, Israel
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oculistica, Rome, Lazio
  - Ospedale Pediatrico Bambino Gesù - Oculistica, Rome, Lazio
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Oculistica, Milan, Lombardy
  - A.O. di Perugia_Hospital Santa Maria della Misericordia - S.C. Oculistica, Perugia, Umbria
- Japan (10):
  - Hospital of the University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Okinawa Prefectural Nanbu Medical Center and Children's MC, Shimajiri-gun, Okinawa
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - Tokyo Metropolitan Ohtsuka Hospital, Toshima-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- Maxima Medisch Centrum, locatie Veldhoven, Veldhoven, Netherlands
- Portugal (2):
  - Hospital Prof. Dr. Fernando Fonseca, Amadora, Lisbon District
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Lisbon
- Romania (2):
  - Clinical Emergency County Hospital, Cluj-Napoca, Cluj
  - Spitalul Clinic de Obstretica si Ginecologie "Cuza Voda", Iași
- Russia (3):
  - FSAI NMRC IRTC "Eye Microsurgery", Kaluga's Branch, Kaluga
  - FGBUZ "NPC of special children care n.a. Voino-Yaseneckogo", Moscow
  - City Children Hospital ?1, Saint Petersburg
- KK Women's and Children's Hospital, Singapore, Singapore
- Narodny ustav detskych chorob, Bratislava, Slovakia
- South Korea (2):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan, Chungcheongnam-do
  - Asan Medical Center - Oncology Department, Seoul, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital la Paz - oftalmologia, Madrid
  - Hospital Universitario Regional De Malaga - Oftalmologia, Málaga
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (5):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Saglik Bilimleri Universitesi Antalya EA Hastanesi, Antalya
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Adana Sehir Egitim ve Arastirma Hastanesi, Yüreğir
- Institute of Eye Diseases and Tissue Therapy named after V.I. Filatov, Consultative Polyclinic, Odesa, Ukraine
- Birmingham Womens Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Stahl A, Nakanishi H, Lepore D, Wu WC, Azuma N, Jacas C, Vitti R, Athanikar A, Chu K, Iveli P, Zhao F, Leal S, Schlief S, Schmelter T, Miller T, Kofuncu E, Fielder A; FIREFLEYE next Study Group. Intravitreal Aflibercept vs Laser Therapy for Retinopathy of Prematurity: Two-Year Efficacy and Safety Outcomes in the Nonrandomized Controlled Trial FIREFLEYE next. JAMA Netw Open. 2024 Apr 1;7(4):e248383. doi: 10.1001/jamanetworkopen.2024.8383. PMID 38687481